CLINICAL TRIAL: NCT03957681
Title: A Phase 3, Placebo-controlled, Double-blind Comparative Study of KHK4827 With an Open-label Extension Period in Subjects With Systemic Sclerosis Who Have Moderate to Severe Skin Thickening
Brief Title: A Phase 3 Study of KHK4827 in Patients With Systemic Sclerosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4827-008
Record Dates: First submitted 2019-05-16; First posted 2019-05-21 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Moderate to Severe Systemic Sclerosis
Keywords: systemic sclerosis; brodalumab; KHK4827
MeSH Terms: conditions — Scleroderma, Systemic | interventions — brodalumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KHK4827 (Experimental)
  Interventions: Drug: KHK4827
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KHK4827 — 210 mg Q2W, SC
  Arms: KHK4827
Drug: Placebo — Q2W, SC
  Arms: Placebo

SUMMARY:
To evaluate the efficacy and safety of KHK4827 in patients with systemic sclerosis who have moderate to severe skin thickening

ELIGIBILITY:
Inclusion Criteria:

* Subject meets the criteria for diagnosis of the Diagnostic Criteria, Severity Classification, and Clinical Practice Guidelines for Systemic Sclerosis （Japanese Dermatological Association 2016） at the pre-examination
* Subject presented the first symptoms of sclerosis other than Raynaud's phenomenon within 60 months before enrollment
* Subject who has systemic sclerosis accompanied by moderate to severe skin thickening with an mRSS of 10 to <30 at the pre-examination and who has progressing skin thickening

Exclusion Criteria:

1. Any of the following significant concomitant diseases:

   * Type 1 diabetes
   * Poorly controlled type 2 diabetes (HbA1c > 8.5%)
   * Congestive heart failure (Class II to IV of the New York Heart Association Functional Classification)
   * Myocartial infarction, unstable angina, or stroke occurring within 12 months before the first dose of investigational product
   * Poorly controlled hypertension (systolic pressure > 150 mm Hg or diastolic pressure > 90 mg Hg at screening)
   * Severe chronic lung disease (%FVC < 60% and %DLco < 40%, calculated according to the Reference Values for Spirometry, Including Viral Capacity, in Japanese Adults Calcluated with the LMS Method and Compared with Previous Values [Japanese Respiratory Society])
   * Major chronic inflammatory diseases or connective tissue diseases other than scleroderma
2. Patient has a history or evidence of a psychiatric disorder, alcohol and/or substance abuse, or any other mental health disorder that, in the opinion of the investigators, would pose a risk to subject safety or interfere with the study evaluation, procedures or completion
3. Patient has a history or evidence of suicidal ideation (severity of 4 or 5) or any suicidal behavior based on an assessment with the Columbia-Suicide Severity Rating Scale (C-SSRS) at enrollment
4. Patient has severe depression based on a total score of ≥ 15 on the Patient Health Questionnaire-8 (PHQ-8) at enrollment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-05-23 (Actual); Primary Completion 2020-10-16 (Actual); Study Completion 2025-04-11 (Actual)

PRIMARY OUTCOMES:
Change in modified Rodnan skin score (mRSS) from baseline at Week 24 | at least 2 weeks up to 24 weeks
  mRSS: scored 0(normal), 1(mild), 2(moderate), or 3(severe) per each site, assessed in 17 different body sites, total score=51

SECONDARY OUTCOMES:
Change in modified Rodnan skin score (mRSS) from baseline at Week 52 | at least 2 weeks up to 52 weeks

CONTACTS AND LOCATIONS:
Locations (6):
- Japan (6):
  - Chukyo Hospital, Nagoya, Aichi-ken
  - The University of Tokyo Hospital, Tokyo, Bunkyo-ku
  - The University of Fukui Hospital, Yoshida-gun, Fukui
  - St. Marianna University School of Medecine Hospital, Kawasaki, Kanagawa
  - Osaka University Hospital, Suita, Osaka
  - Fukushima Medical University Hospital, Fukushima

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make IPD and related data dictionaries available. The datasets generated and/or analyzed during the study sponsored by Kyowa Kirin will be available in the Vivli repository, https://vivli.org/ourmember/kyowa-kirin/ as long as conditions of data disclosure specified in the policy section of the Vivli website are satisfied.
URL: https://vivli.org/ourmember/kyowa-kirin/